CLINICAL TRIAL: NCT05904444
Title: The Effect of Duration Between Sessions on Microperimetric Biofeedback Training in Patients With Maculopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aier Eye Hospital, Guangzhou (Other)
Responsible Party: Principal Investigator, Jie Zhou, Resident doctor, Aier Eye Hospital, Guangzhou
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZAIER2018IRB11
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Macular Degeneration; Low Vision; Stargardt Disease
Keywords: Macular disease; low vision; Visual rehabilitation
MeSH Terms: conditions — Macular Degeneration; Vision, Low; Stargardt Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- daily training (Experimental): Patients underwent microperimetric training on everyday
  Interventions: Procedure: microperimetric biofeedback training
- alternately training (Experimental): Patients underwent microperimetric training on every other day
  Interventions: Procedure: microperimetric biofeedback training

INTERVENTIONS:
Procedure: microperimetric biofeedback training — Microperimetry biofeedback training is a noninvasive stragegy to develop a new trained retinal locus or strength the spontaneous preferred retinal locus to get better visual performances.The rationale of MBFT consists in reeducating visual system to a new visual condition, promoting retina-brain transmission, and further enhancing synaptic plasticity and neural capacity by acoustic biofeedback or structured light stimulus biofeedback.

SUMMARY:
Patients who develop macular diseases have several clinical complications,such as central vision loss, the central scotoma of the visual field, the decrease of reading speed and fixation stability. At present, there is still no satisfactory effect in the prevention and treatment of advanced macular disease. A new rehabitation strategy named microperimetric biofeedback training has been shown to be effective in improving patients' visual appearance, but there is no consensus regarding the optimal methodology and standard of practice. Therefore, we designed a prospective clinical study to verify the effectiveness of MBFT and to determine an optimal plan.

DETAILED DESCRIPTION:
The present study aimed to investigate the effects of training frequency and number of training sessions on the visual outcomes of patients with various macular diseases. A total of 15 training sessions were conducted on two distinct frequencies, namely once a day and once every other day. Baseline measurements included fixation stability, reading speed, and best corrected visual acuity (BCVA) were obtained and followed up after the 5, 10, and 15 training sessions. By comparing the changes in these visual function parameters across different stages of training, the study aimed to identify and analyze the underlying patterns and rules governing the training process. Ultimately, the results of this study could serve as a valuable reference for standardizing the use of MBFT in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

participants who (1) were diagnosed with macular disease and had a BCVA poorer than 20/60; (2) with stable fundus lesion in fundus examinations; (3)with education level beyond the third grade; (4)had no other effective treatment; and (5)were willing to improve visual quality.

Exclusion Criteria:

who (1) received ocular treatments in the preceding 3 months, (2) with active fundus lesions like inflammation, bleeding, exudation, edema, (3) with obvious opacity of the refractive media such as keratopathy, severe cataract, or severe vitreous opacity, (4) were unable to attend scheduled follow-up appointments.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
fixation stability | 5 minutes
  An index for evaluating macular disease, defined as the accuracy of a patient's gaze at a target over a period of time.

SECONDARY OUTCOMES:
Best corrected visual acuity | 2 minutes
  The most important indicator of visual function, refers to the function of distinguishing objects in the state of refractive correction.
Reading speed | 3 minutes
  One of the indicators for evaluating reading ability, which refers to the number of words within a certain period of time when reading
Questionnaires | 10 minutes
  Questionnaires were used to determine the influence of eye symptoms and visual impairment on daily life attributed to the limitation of patients' social function and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jinling Zhang, doctor, Study Director — Aier Eye Hospital, Guangzhou
Locations (1):
- MAIA microperimetry, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Maniglia M, Visscher KM, Seitz AR. Perspective on Vision Science-Informed Interventions for Central Vision Loss. Front Neurosci. 2021 Nov 4;15:734970. doi: 10.3389/fnins.2021.734970. eCollection 2021. PMID 34803584
- [Result] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Result] Wang Y, Ye J, Shen M, Yao A, Xue A, Fan Y, Huang S, Wang J, Lu F, Shao Y. Photoreceptor Degeneration is Correlated With the Deterioration of Macular Retinal Sensitivity in High Myopia. Invest Ophthalmol Vis Sci. 2019 Jul 1;60(8):2800-2810. doi: 10.1167/iovs.18-26085. PMID 31266057
- [Result] Fletcher DC, Schuchard RA. Preferred retinal loci relationship to macular scotomas in a low-vision population. Ophthalmology. 1997 Apr;104(4):632-8. doi: 10.1016/s0161-6420(97)30260-7. PMID 9111255
- [Result] Maniglia M, Soler V, Cottereau B, Trotter Y. Spontaneous and training-induced cortical plasticity in MD patients: Hints from lateral masking. Sci Rep. 2018 Jan 8;8(1):90. doi: 10.1038/s41598-017-18261-6. PMID 29311565
- [Result] Vingolo EM, Napolitano G, Fragiotta S. Microperimetric biofeedback training: fundamentals, strategies and perspectives. Front Biosci (Schol Ed). 2018 Jan 1;10(1):48-64. doi: 10.2741/s500. PMID 28930518
- [Result] Morales MU, Saker S, Wilde C, Rubinstein M, Limoli P, Amoaku WM. Biofeedback fixation training method for improving eccentric vision in patients with loss of foveal function secondary to different maculopathies. Int Ophthalmol. 2020 Feb;40(2):305-312. doi: 10.1007/s10792-019-01180-y. Epub 2019 Oct 3. PMID 31583549
- [Result] Sahli E, Altinbay D, Bingol Kiziltunc P, Idil A. Effectiveness of Low Vision Rehabilitation Using Microperimetric Acoustic Biofeedback Training in Patients with Central Scotoma. Curr Eye Res. 2021 May;46(5):731-738. doi: 10.1080/02713683.2020.1833348. Epub 2020 Oct 18. PMID 33073619
- [Result] Raman R, Damkondwar D, Neriyanuri S, Sharma T. Microperimetry biofeedback training in a patient with bilateral myopic macular degeneration with central scotoma. Indian J Ophthalmol. 2015 Jun;63(6):534-6. doi: 10.4103/0301-4738.162609. PMID 26265646
- [Result] Bozkurt Oflaz A, Turgut Ozturk B, Gonul S, Bakbak B, Gedik S, Okudan S. Short-Term Clinical Results of Preferred Retinal Locus Training. Turk J Ophthalmol. 2022 Feb 23;52(1):14-22. doi: 10.4274/tjo.galenos.2021.73368. PMID 35196835